CLINICAL TRIAL: NCT01023828
Title: K-RAS Oncogene Mutation in Patients With Advanced Non-Small Cell Lung Cancer Associated With Exposure to Wood Smoke and Tobacco Smoking: Therapeutic Implications
Acronym: 007/055/OMI
Status: Completed | Type: Observational
Sponsor: National Institute of Cancerología (Other Government)
Collaborators: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, DR. MYRNA CANDELARIA, MD, National Institute of Cancerología
Other Study IDs: INCAN/CC/394/07
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: K-RAS ONCOGENE MUTATION; NON-SMALL CELL LUNG CANCER; WOOD SMOKE
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The tumor samples, both formalin-fixed or paraffin-embedded, used for the histological diagnosis of patients will be obtained from the Pathology Departments of the National Cancer Institute and the National Institute of Respiratory Diseases; these samples will be used to gather DNA for the analysis of K-RAS mutations. The clinical data of the patients will be obtained from their medical files.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- TOBACCO SMOKING: Group of patients with diagnosis of NSCLC and exposure to tabacco smoking
- WOOD SMOKE: Patients whit diagnosis of NSCLC and exposure to wood smoke
- TABACCO SMOKING AND WOOD SMOKE: Patients whit diagnosis of NSCLC and exposure to tabacco smoking and wood smoke
- WHITOUT EXPOSURE: Patients whit diagnosis of NSCLC and whitout exposure to risk factor

SUMMARY:
Summary:

Non-small cell lung cancer (NSCLC) is the leading cause of cancer-related death in the world. This neoplasia has a poor survival prognosis due to the low effectiveness of existing treatments. The low effectiveness is associated with the development of an intrinsic and acquired resistance of tumors, which clinically shows through early progression and transitory responses. Tobacco smoking is the major risk factor for NSCLC; however, wood smoke has been described as a strong carcinogen and a relevant risk factor for the development of NSCLC. Current data indicates that lung tumors associated with tobacco smoking and wood smoke show different clinical characteristics, which suggests that they might also have different genetic alterations, which are a consequence of tumor etiology. The description of the frequency and the type of mutations associated with different etiologies of NSCLC could represent the starting point for benefiting each patient according to their specific characteristics. One of the most researched signaling pathways related to cancer cell proliferation is the one activated by the K-RAS oncogene. Active K-RAS mutations have been detected in different types of neoplasia and more than 90% of these mutations occur at codon 12 of the oncogene. These mutations seem to be an independent risk factor for the prognosis of malignant tumors and they are associated with the lack of response to erlotinib, which is a tyrosine-kinase inhibitor. The investigators' research team has recently reported that wood smoke is an independent factor for survival and response to the erlotinib treatment, which suggests that this carcinogen could have a different frequency and pattern of mutations in the K-RAS oncogene, compared to what has been reported in smoking patients. Determining the tumor mutations within the K-RAS oncogene can help improve the response prognosis of patients with advanced NSCLC who have a background of exposure to different factors associated with the appearance of this neoplasia, such as wood smoke exposure or tobacco smoking. Therefore, the objective of this research is to determine the frequency and the type of mutations at codon 12 of the K-RAS oncogene in patients with NSCLC who have a background of exposure to tobacco smoking or wood smoke.

DETAILED DESCRIPTION:
Background:

Lung cancer is the leading cause of cancer-related death among men and women worldwide (1). In 2007, 213,380 new cases of lung cancer were registered; from these cases, 160,390 deaths were reported. This number represents 15% of the total cases and 29% of cancer-related deaths in the world. Only 13% of the patients with lung cancer survive for 5 years [surveillance epidemiology and end result (seer) statistics http://seer. cancer.gov/], therefore it still is a serious health problem (2). Clinically speaking, lung cancer is divided into two main categories that cover small cell lung cancer and non-small cell lung cancer (NSCLC). About 75% of all lung tumors are NSCLC, including squamous cell carcinoma, adenocarcinoma, and large cell carcinoma (1). Despite the multimodal treatment using chemotherapy, radiotherapy and surgery there is a poor prognosis for locally advanced NSCLC. Survival rates for clinical stage IIIA is 64% at one year and between 23% and 30% after five years; for clinical stage IIIB 32% and 3% after one and five years, respectively (3). While advancements in the treatment of NSCLC have been made, few survival rate improvements have been achieved.

Tobacco smoking is considered the main cause of NSCLC, but there are other risk factors as well, such as the exposure to asbestos, radon, heavy metals, and wood smoke. The latter has been described as a human carcinogen and an important risk factor for the development of NSCLC. The frequency of exposure to wood smoke in patients with NSCLC is 28% (2). Current data indicates than lung cancer associated with tobacco smoking and the lung cancer associated with wood smoke exposure present different clinical characteristics, which suggests that they might also have different genetic alterations, which are a consequence of tumor etiology. Nevertheless, there are no significant molecular researches that make possible to determine the differences in the pattern of mutations in oncogenes involved in lung tumorigenesis, in relation to the risk factors accounted by the patient. Recent advances in the knowledge of cancer biology have led to the identification of various potential molecular targets that play a major role in the development and progression of the disease. One of the most extensively researched signaling pathways involved in the cell proliferation and survival is the one activated by the epidermal growth factor receptor (EGFR). When the epidermal growth factor (EGF) binds to the extracellular domain of EGFR the kinase property of the receptor is activated regulating the activation of different signaling pathways. One of these pathways leads to the activation of K-RAS, which at the same time activates the pathway of MAP kinase, involved in the proliferation, differentiation, migration, and survival of the cell (these are fundamental events in oncogenesis). Reports indicate that mutations in EGFR can be found in 51% of non-smoking patients (4) and in 10% of smoking patients, while mutations in K-RAS occur in 30% to 50% of the lung adenocarcinomas associated with tobacco.

Active mutations in K-RAS not only occur in NSCLC, but they also occur in >50% of the colorectal adenocarcinomas, 75% of pancreatic tumors, 48% of lung cancer, and 44% of adrenocortical tumors (5). These mutations seem to be an independent risk factor for the prognosis of malignant tumors, since more than 90% of them occur at the codon 12 of the K-RAS gene (6-8), and they are associated with lack of response to erlotinib (9), a tyrosine-kinase inhibitor. Our research team has recently reported that wood smoke is an independent factor for the survival and response to a treatment with erlotinib (10). This information strongly supports the hypothesis that lung cancer tumorigenesis results from different molecular mechanisms according to the smoker's stage (11) or other carcinogenic factors associated with the appearance of the malignant neoplasia, such as wood smoke exposure. Therefore, we believe that, compared to what has been reported in smoking patients, wood smoke could cause a different frequency and pattern of mutations in the K-RAS oncogene. It is of clinical relevance to determine whether the patients with NSCLC exposed to wood smoke present any differences in the frequency and the type of mutations in the K-RAS gene, with respect to both smoking and non-smoking patients.

Actually, a number of potential biological markers are being investigated with the aim of selecting patients who will receive more specific therapies and thus achieve better results regarding the response to treatment and overall survival. This is why the ability to detect K-RAS mutations associated with risk factors for NSCLC could represent a starting point for proposing different treatment approaches and benefiting the patients according to the specific characteristics of each tumor.

General Objective:

To define the frequency and type of mutations at codon 12 of the K-RAS oncogene that occur in patients with non-small cell lung cancer who have a background of wood smoke exposure or tobacco smoking.

Materials and Methods:

The presence of mutations at the K-RAS oncogene will be evaluated retrospectively in 50 patients with advanced NSCLC who have a background of wood smoke exposure and 50 patients with NSCLC who have a background of tobacco smoking. Additionally, 50 patients with NSCLC with or without a background of exposure to any of these risk factors for lung cancer will be prospectively evaluated. For the patients that will be prospectively studied, the inclusion criteria will be as follows: patients diagnosed with advanced NSCLC stage IIIB/IV who have not received previous chemotherapy, radiotherapy or both and who have tumor tissue embedded in paraffin blocks or formalin-fixed; these patients must sign an informed consent letter. The exclusion criteria will be: patients who refuse to participate in the study or those who decide to withdraw from it, patients without tumor tissue or with a poor quality sample. The tumor samples, both formalin-fixed or paraffin-embedded, used for the histological diagnosis of patients will be obtained from the Pathology Departments of the National Cancer Institute and the National Institute of Respiratory Diseases; these samples will be used to gather DNA for the analysis of K-RAS mutations. The clinical data of the patients will be obtained from their medical files.

DNA extraction:

Genomic DNA was extracted by standard procedure from areas of paraffin slides containing >50% tumor using the QIAamp DNAFFPE Tissue Kit (QIAGEN), according to the manufacturer's instructions.

Analysis of K-RAS oncogene mutations KRAS gene mutations from the samples were detected by Therascreen RGQ PCR Kit (QUIAGEN, Scorpions ARMS method), according to the manufacturer's instructions.

For the statistical analysis of results, continuous variables will be presented as arithmetic means, medians, and standard deviations, while the categorical variables will be presented as proportions and 95% confidence intervals. Inferential comparisons will be performed by Student's t test and Mann-Whitney U test, according to the distribution of data (normal and abnormal) determined by the Kolmogorov-Smirnov test. Either the chi square test or the Fisher's exact test will be performed to evaluate significance among categorical variables. Statistic significance will be determined as a p<0.05 value with a two- tailed test. Both significant variables and variables with a borderline significance (p<0.1) will be included in the multivariate logistic regression analysis. Comparisons between groups will be carried out with the log-rank test.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with advanced NSCLC stage IIIB/IV who have not received previous chemotherapy
* Radiotherapy or both and who have tumor tissue embedded in paraffin blocks or formalin-fixed
* These patients must sign an informed consent letter.

Exclusion Criteria:

* Patients who refuse to participate in the study or those who decide to withdraw from it.
* Patients without tumor tissue or with a poor quality sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For the purpose of this research, the presence of mutations at the K-RAS oncogene were evaluated retrospectively in 50 patients with advanced NSCLC who have a background of wood smoke exposure and 50 patients with NSCLC who have a background of tobacco smoking. Additionally, 50 patients with NSCLC with or without a background of exposure to any of these risk factors for lung cancer will be prospectively evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2005-04; Primary Completion 2010-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
History of smoking and wood smoke exposure | Exposure factor
  Tumor specimens were collected at the time of diagnosis. WSE was defined as being exposed to fumes resulting from burning wood in fireplaces and wood stoves for >5 years for at least 4 hours per day. The WSE index was calculated by multiplying the number of daily hours exposed by the number of years' exposure. A non-smoker was defined as being someone having a lifetime exposure of less than 100 cigarettes; the tobacco smoking index was calculated by multiplying the number of cigarette packs consumed per day by the number of years spent smoking.

SECONDARY OUTCOMES:
KRAS and EGFR mutations | Genotyping
  EGFR (exon 18-21) and KRAS gene mutations from some samples were detected by Therascreen RGQ PCR Kit (QUIAGEN, Scorpions ARMS method), according to the manufacturer's instructions from the four arms.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD; MsC, Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- Instituto Nacional de Cancerología, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Campos-Parra AD, Aviles A, Contreras-Reyes S, Rojas-Marin CE, Sanchez-Reyes R, Borbolla-Escoboza RJ, Arrieta O. Relevance of the novel IASLC/ATS/ERS classification of lung adenocarcinoma in advanced disease. Eur Respir J. 2014 May;43(5):1439-47. doi: 10.1183/09031936.00138813. Epub 2014 Jan 16. PMID 24435003
- [Derived] Campos-Parra AD, Zuloaga C, Manriquez ME, Aviles A, Borbolla-Escoboza J, Cardona A, Meneses A, Arrieta O. KRAS mutation as the biomarker of response to chemotherapy and EGFR-TKIs in patients with advanced non-small cell lung cancer: clues for its potential use in second-line therapy decision making. Am J Clin Oncol. 2015 Feb;38(1):33-40. doi: 10.1097/COC.0b013e318287bb23. PMID 23538866
- [Derived] Arrieta O, Campos-Parra AD, Zuloaga C, Aviles A, Sanchez-Reyes R, Manriquez ME, Covian-Molina E, Martinez-Barrera L, Meneses A, Cardona A, Borbolla-Escoboza JR. Clinical and pathological characteristics, outcome and mutational profiles regarding non-small-cell lung cancer related to wood-smoke exposure. J Thorac Oncol. 2012 Aug;7(8):1228-34. doi: 10.1097/JTO.0b013e3182582a93. PMID 22659961